CLINICAL TRIAL: NCT00701558
Title: An Open Label Study to Evaluate the Effect of First Line Treatment With Tarceva in Combination With Gemcitabine on Disease Progression in Patients With Unresectable Advanced and/or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of First Line Treatment With Tarceva (Erlotinib) in Combination With Gemcitabine in Patients With Unresectable Advanced and/or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20951; 2007-002135-83
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Erlotinib Hydrochloride; Gemcitabine

ARMS (1):
- Erlotinib + Gemcitabine (Experimental): Participants received erlotinib 150 mg/day, orally (po) on a continuous schedule in combination with gemcitabine at 1000 mg/m^2 administered intravenously (iv) on days 1, 8, 15 of each 4 week cycle for 6 cycles as per standard medical care, or until disease progression or participant's withdrawal due to any reason or death.
  Interventions: Drug: Erlotinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Erlotinib — 150 mg po daily
  Other Names: Tarceva
Drug: Gemcitabine — 1000 mg/m^2 iv on days 1, 8, 15 of each 4 week cycle for 6 cycles

SUMMARY:
This single arm study will assess the efficacy and safety of erlotinib + gemcitabine in chemotherapy-naive participants with unresectable, advanced and/or metastatic non-small cell lung cancer. Participants will receive erlotinib 150 mg orally (po) daily, in combination with gemcitabine 1000 mg/m^2 intravenously (iv) weekly for 3 weeks of each 4 week cycle. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* advanced and/or metastatic (stage IIIB/IV) unresectable non-small cell lung cancer;
* no previous systemic chemotherapy, radiation therapy or immunotherapy;
* Eastern Cooperative Oncology Group (ECOG) >=2.

Exclusion Criteria:

* prior systemic anti-tumor therapy with human epidermal growth factor receptor 1 (HER1/EGFR) inhibitors;
* active, non-controlled systemic disease;
* any other malignancies within 5 years (except for adequately treated cancer in situ of cervix, or basal or squamous cell skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib + Gemcitabine
Started | 19
Completed | 4
Not Completed | 15
Not completed — Death | 7
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.47 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Time to disease progression or progression free survival (PFS) was defined as the interval between the day of randomization and the date of the first documentation of disease progression or date of death (from any cause), whichever occurs first.
Time Frame: From the time of randomization until disease progression or death (up to 193 weeks)]
Population: Intention to treat (ITT) population included all participants who were randomized to treatment group.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 18
weeks | 15 [7 to 36]

2. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the percentage of participants who had any evidence of confirmed objective complete response (CR) or partial response (PR), per the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) and assessed by computed tomography imaging (CT): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the time of randomization until disease progression or death (up to 193 weeks)
Population: ITT population included all participants who were randomized to treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 19
percentage of participants | 15.8

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval between the day of randomization and the date of death from any cause.
Time Frame: From the time of randomization until death (up to 193 weeks)
Population: ITT population included all participants who were randomized to treatment group.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 19
weeks | 39 [27 to 51]

ADVERSE EVENTS:
Time Frame: Up to 28 days after last study drug administration in the study treatment phase (up to 197 Weeks)
Arm/Group | Erlotinib + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Gemcitabine (N=19)
Diarrhoea (Gastrointestinal disorders) | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Gemcitabine (N=19)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Blood bilirubin increased (Investigations) | 2
Appetite lost (Metabolism and nutrition disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights